CLINICAL TRIAL: NCT04561856
Title: Fascia Iliaca Block Supplemented With Perineural Vs Intravenous Dexamethasone: Effect On Post-Operative Pain In Children Undergoing Split Thickness Skin Grafting.
Brief Title: Fascia Iliaca Block Supplemented With Perineural Vs Intravenous Dexamethasone
Acronym: Interventional
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mahmoud Abbas, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIBS
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1 (Active Comparator): will include 33 patients: each one will receive US guided fascia-iliaca block with 0.7 ml/kg of bupivacaine 0.25% plus 2 ml of normal saline perinural plus 0.15 mg/kg dexamethasone (maximum of 4 mg) in 2 ml volume intravenously.
  Interventions: Drug: Dexamethasone
- Group2 (Active Comparator): will include 33 patients: each one will receive US guided fascia-iliaca block with 0.7 ml/kg of bupivacaine 0.25% plus 0.15 mg/kg dexamethasone (maximum of 4 mg) in 2 ml volume perinural plus 2 ml of normal saline intravenously.
  Interventions: Drug: Dexamethasone
- Group3 (Placebo Comparator): will include 33 patients: each one will receive US guided fascia-iliaca block with 0.7 ml/kg of bupivacaine 0.25% plus 2 ml of normal saline perinural plus 2 ml of normal saline intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Intravenous 4mg
  Arms: Group1
Drug: Dexamethasone — Perineural 4mg
  Arms: Group2
Drug: Placebo — Normal Saline 2ml
  Arms: Group3

SUMMARY:
Split-thickness skin grafting is the current standard of care for the reconstructive procedures in managing burn injuries and traumatic tissue defects. Harvesting split-thickness skin creates a new partial thickness wound that is referred to as the donor site . Donor site pain is one of the most distressing symptoms reported by patients in the early postoperative period. Larger donor sites stimulate a greater number of pain receptors and consequently pain is proportional to the size of the graft harvested.Often, the donor site is reported to be more painful than the recipient site,affecting early mobilization, sleep, and need for analgesics postoperatively.

DETAILED DESCRIPTION:
Most commonly split thickness auto-grafts are harvested from a convenient and minimally aesthetically intrusive site; often the lateral thigh area, which is innervated by lateral femoral cutaneous nerve (LFCN). However if a larger graft area in needed then it will be obtained from the anterior aspect of the thigh, which is innervated by the femoral nerve.

Regional nerve blockade has been proposed for skin graft harvest and proofed to provide better and longer standing analgesia. Application of fascia iliaca compartment block involves the distribution of anesthesia to the territories of the femoral and lateral cutaneous nerves.

American society of regional anesthesia and pain medicine recommendations on local anesthetics in pediatric regional anesthesia in 2018 stated that the ultrasound guided fascial plane blocks as fascia iliaca block can be successfully and safely performed using a recommended dose of 0.25-0.75 mg/kg of bupivacaine 0.25%.

Prolongation of analgesia after surgery under regional anaesthesia is a goal for clinicians. Many investigators have sought that the ideal analgesic adjuvant that would both prolongs pain relief and avoids side effects after a single-shot peripheral nerve block. Although many agents have failed this test (opioids, ketamine, clonidine, etc.), the perineural addition of dexamethasone to local anaesthetic has been shown in several studies to prolong the analgesic effect and its use has become common in clinical practice around the world. Not surprisingly, much research has been performed with the aim of providing Level 1 evidence via randomized controlled trials design and systematic review and meta-analysis. Despite this, there is still no adequate answer as to whether perineural dexamethasone is superior to systemic administration alone.

ELIGIBILITY:
Inclusion Criteria: • Age 2 -12 years.

* ASA I - II
* Scheduled for split thickness grafting.
* Availability and suitability of lateral and anterior aspects of the thigh as a donor site.

Exclusion Criteria:

* Patient's guardian refusal to participate in the study.
* Known allergy to local anesthetics
* Children known to be diabetic.
* Coagulopathy.
* Children with motor or sensory deficits in lower extremities.
* Children who are morbidly obese (BMI≥35) because ultrasound guided regional anesthesia could be technically difficult.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Time of first postoperative analgesia requirement using FLACC score | 24 Hours
  FLACC Score for the first 24 hours postoperative; 0 = Relaxed and comfortable, 1-3 = Mild discomfort, 4-6 = Moderate pain, 7-10 = Severe discomfort/pain or both.And The total consumption of postoperative rescue analgesics (total of paracetamol doses) will be recorded over 24 hours.

SECONDARY OUTCOMES:
Intraoperative blood pressure | 24 Hours
  Intraoperative blood pressure will be recorded every 3 minutes till the end of the procedure then postoperative at 1,2, 4,8,12,16 and 24 hours.
Intraoperative heart rate | 24 Hours
  Intraoperative heart rate will be recorded every 3 minutes till the end of the procedure then postoperative at 1,2, 4,8,12,16 and 24 hours.

REFERENCES:
- [Result] Sinha S, Schreiner AJ, Biernaskie J, Nickerson D, Gabriel VA. Treating pain on skin graft donor sites: Review and clinical recommendations. J Trauma Acute Care Surg. 2017 Nov;83(5):954-964. doi: 10.1097/TA.0000000000001615. PMID 28598907
- [Result] Shank ES, Martyn JA, Donelan MB, Perrone A, Firth PG, Driscoll DN. Ultrasound-Guided Regional Anesthesia for Pediatric Burn Reconstructive Surgery: A Prospective Study. J Burn Care Res. 2016 May-Jun;37(3):e213-7. doi: 10.1097/BCR.0000000000000174. PMID 25412051
- [Result] Shteynberg A, Riina LH, Glickman LT, Meringolo JN, Simpson RL. Ultrasound guided lateral femoral cutaneous nerve (LFCN) block: safe and simple anesthesia for harvesting skin grafts. Burns. 2013 Feb;39(1):146-9. doi: 10.1016/j.burns.2012.02.015. Epub 2012 May 30. PMID 22657583
- [Result] Suresh S, Ecoffey C, Bosenberg A, Lonnqvist PA, de Oliveira GS Jr, de Leon Casasola O, de Andres J, Ivani G. The European Society of Regional Anaesthesia and Pain Therapy/American Society of Regional Anesthesia and Pain Medicine Recommendations on Local Anesthetics and Adjuvants Dosage in Pediatric Regional Anesthesia. Reg Anesth Pain Med. 2018 Feb;43(2):211-216. doi: 10.1097/AAP.0000000000000702. PMID 29319604
- [Result] Hewson D, Bedforth N, McCartney C, Hardman J. Dexamethasone and peripheral nerve blocks: back to basic (science). Br J Anaesth. 2019 Apr;122(4):411-412. doi: 10.1016/j.bja.2019.02.004. Epub 2019 Feb 25. No abstract available. PMID 30857596
- [Result] Veneziano G, Martin DP, Beltran R, Barry N, Tumin D, Burrier C, Klingele K, Bhalla T, Tobias JD. Dexamethasone as an Adjuvant to Femoral Nerve Block in Children and Adolescents Undergoing Knee Arthroscopy: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial. Reg Anesth Pain Med. 2018 May;43(4):438-444. doi: 10.1097/AAP.0000000000000739. PMID 29377866